CLINICAL TRIAL: NCT05327998
Title: Pilot Study of Renal Function by a Reference Isotopic Technique in Malnourished Patients With Anorexia Nervosa
Brief Title: Kidney Function and Anorexia Nervosa
Acronym: ANKID
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211173; 2021-A01538-33 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa; Kidney Injury
Keywords: anorexia nervosa; renal function; undernutrition; eating disorder; glomerular filtration rate (GFR); cystatin C
MeSH Terms: conditions — Anorexia Nervosa; Malnutrition; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anorexia nervosa (AN) is an eating disorder that can lead to severe medical complications. Kidney injuries are unknown in patients with extremely malnourished AN (BMI <13). The primary objective of the study is to evaluate the frequency and to determine the profiles of patients who may develop kidney injuries. The secondary objective is to evaluate the evolution of kidney injuries after a phase of refeeding. Guidelines for medical treatments and dietary intakes will be recommended to avoid severe or irreversible renal disease.

DETAILED DESCRIPTION:
Anorexia nervosa is an eating disorder that can lead to undernutrition and severe somatic complications. The clinical nutrition unit in Paul Brousse hospital provide care to adult patients with a severe forms of AN. Kidney complications are poorly known and little explored. Indeed, patients suffering from AN have a higher prevalence of kidney failure due to the absence of a reference methods. Kidney injuries come from multiple origin like chronic ionic disorders, dehydration and hyperprotein diet. The aim of this study will be to evaluate kidney injuries and to follow its evolution during refeeding. Blood and urine simple of Cystatine C will be add to routine analyses. This will allow us to know if, there is a concordance between the reference technique (measurement of glomerular filtration rate by isotopic method 99mTC-DTPA) and the measurement of Cystatin C. Thus, guidelines of dietary intake and medical treatments can be achieved in order to prevent severe forms requiring dialysis and kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with undernutrition (BMI < 18,5);
* Patient with AN according to DSM-5 criteria, validated by Eating Disorder Diagnostic Scale and EDDS-questionnaire;
* Patient informed and signed a consent form;
* Patient affiliated to a social security plan.

Exclusion Criteria:

* Patient no-reponding to all criteria of DSM-5;
* Patient with a renal comorbidity no-related to AN;
* Patient under AME scheme;
* Pregnancy or breastfeeding;
* Participation to another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anorexia nervosa
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
DFG measurement | at 18 months
  Measurement of glomerular filtration rate by 99mTc-DTPA isotopic technic.
  Glomerular Filtration Rate (GFR) measurement by isotopic technique remains the best quantitative marker of kidney function. It allows the diagnosis and the classification of the severity of chronic kidney disease into five stages. Several methods and radiopharmaceutical markers have been developed. The main radiopharmaceuticals used are technetium-labeled diethylene-triamino-penta-acetate (99mTC-DTPA), iodine-labeled iothalamate (125I-iothalamate), and chromium-51-labeled ethylenediaminetetraacetic acid (I51Cr-EDTA). The main advantages of these compounds are : high assay accuracy and a rapid distribution. They can be used in urinary and plasma clearance alternatively. The limitations regarding radioactive products, even if the irradiation remains very low (4% of the dose received during a thoracic radiography).

SECONDARY OUTCOMES:
Cystatin C and predictive formulas for measuring GFR from blood creatinine level | at 18 months
  Cystatin C is secreted by all cell nuclei in the body, filtered by the glomeruli and catabolized in the proximal tubule. Its concentration in the blood is independent of muscle mass. Its level would be better correlated to glomerular filtration measured by 51Cr-EDTA.

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Hanachi, MD, Principal Investigator — Department of Nutrition, Paul Brousse hospital, APHP; Marika Dicembre, Master's, Study Director — Department of Nutrition, Paul Brousse hospital, APHP
Locations (1):
- Department of Nutrition, Paul Brousse hospital, APHP, Villejuif, France

IPD SHARING:
Plan to Share IPD: No